CLINICAL TRIAL: NCT00676689
Title: Implantation of the SAPIEN Transcatheter Heart Valve (THV) in the Pulmonic Position
Brief Title: COMPASSION - COngenital Multicenter Trial of Pulmonic VAlve Regurgitation Studying the SAPIEN InterventIONal THV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-09
Record Dates: First submitted 2008-05-09; First posted 2008-05-13 (Estimated); Results first posted 2016-09-01 (Estimated); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Pulmonary Valve Insufficiency; Pulmonary Regurgitation; Dysfunctional RVOT Conduit; Pulmonary Obstruction; Pulmonary Stenosis
Keywords: Pulmonic; Regurgitation; Pulmonary Valve Conduit; Stenosis; Congenital Heart Defect
MeSH Terms: conditions — Pulmonary Valve Insufficiency; Airway Obstruction; Pulmonary Valve Stenosis; Gastroesophageal Reflux; Constriction, Pathologic; Heart Defects, Congenital

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- SAPIEN THV (Experimental)
  Interventions: Device: SAPIEN Transcatheter Valve Implantation

INTERVENTIONS:
Device: SAPIEN Transcatheter Valve Implantation — Device Implantation

SUMMARY:
To assess the safety and effectiveness of pulmonic THV implantation in subjects with dysfunctional RVOT conduit requiring treatment for moderate or severe pulmonary regurgitation (≥3+ pulmonary regurgitation) and/or RVOT conduit obstruction (mean gradient of >=35mmHg) by TTE.

DETAILED DESCRIPTION:
The study design is a multi-center, prospective, non-randomized study of up to 70 implanted subjects (US) with no site representing more than 30% of the implanted subjects. The subjects will include those subjects who have previously undergone placement of a conduit between the right ventricle and pulmonary artery and now present with a dysfunctional RVOT conduit requiring treatment for moderate or severe pulmonary regurgitation and/or RVOT conduit obstruction.

ELIGIBILITY:
Inclusion Criteria

1. Weight must be equal to or exceed 35 kilograms.
2. In situ conduit size of ≥ 16 mm and ≤ 24 mm in diameter.
3. Subject presents with moderate or severe pulmonary regurgitation defined as ≥3+ pulmonary regurgitation by TTE or RVOT conduit obstruction with a mean gradient of >= 35 mmHg by TTE.
4. Subject is symptomatic as evidenced by cardiopulmonary exercise testing.
5. The subject or the subject's legal representative has been informed of the nature of the study, agrees to its provisions and has provided written informed consent as approved by the Institutional Review Board (IRB) of the respective clinical site.
6. The subject and the treating physician agree that the subject will return for all required post-procedure follow up visits and the subject will comply with protocol-required follow-up visits.
7. Catheterization is determined to be feasible by the treating physician.

Exclusion Criteria

1. Active infection requiring current antibiotic therapy (if temporary illness, subject may be a candidate 4 weeks after discontinuation of antibiotics)
2. Previously enrolled in this study.
3. Subject with pre-existing prosthetic heart valves in any position*.
4. Severe chest wall deformity.
5. Leukopenia (WBC<3000 mm3).
6. Acute or chronic anemia (Hb <9 g/dL).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2008-04-08 (Actual); Primary Completion 2015-11 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ziyad M Hijazi, M.D., Principal Investigator — Rush University Medical Center
Locations (7):
- United States (7):
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Miami Children's Hospital, Miami, Florida
  - Emory University Hospital/ Children's Healthcare of Atlanta (CHOA), Atlanta, Georgia
  - Rush Medical Center, Chicago, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - Children's Hospital of New York, New York, New York
  - Duke University Medical Center, Durham, North Carolina

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SAPIEN THV
Started | 81
Procedure | 79 (Two enrolled patients did not meet eligibility criteria and did not undergo the study procedure.)
30 Day Follow-up | 78
1 Year Follow-up | 64
Completed | 20
Not Completed | 61
Not completed — Screen Failure | 2
Not completed — Death | 2
Not completed — Lost to Follow-up | 4
Not completed — Physician Decision | 1
Not completed — Withdrawal by Subject | 3
Not completed — Continuing FU | 49

BASELINE CHARACTERISTICS:
Population: Safety Population (SP): All enrolled subjects for whom the procedure has begun, regardless of whether the valve was successfully implanted. The definition of "procedure has begun" is "the time of the creation of vascular access - incision or puncture."
Arm/Group | SAPIEN THV
Number analyzed (Participants) | 79
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.0 (13.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 52
New York Heart Association Group [Number; unit: participants] — Class Patient Symptoms I No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation, shortness of breath.
  II Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, shortness of breath.
  III Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, or dyspnea.
  IV Unable to carry on any physical activity without discomfort. Symptoms of heart failure at rest. If any physical activity is undertaken, discomfort increases.
  participants
    Class I/II | 54
    Class III/IV | 25
Primary Indication [Number; unit: participants]
  Pulmonary Stenosis | 7
  Pulmonary Regurgitation | 10
  Both | 62

OUTCOME MEASURES:

1. Primary Outcome: Freedom From Device or Procedure Related Death or Reintervention
Time Frame: 1 year
Population: Valve implant population. There were 2 screen failure patients and 10 patients where the procedure was started but the study valve not implanted, leaving 69 patients in the Valve Implant Population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SAPIEN THV
Number analyzed (Participants) | 69
percentage of participants | 97.1 [88.9 to 99.3]
Statistical Analysis 1: Comparison: SAPIEN THV; Test type: Superiority or Other; Kaplan-Meier = 0.971, 95% CI 2-sided [0.889 to 0.993], Standard Error of Mean 0.020

2. Secondary Outcome: Freedom From MACCE
Description: Clinical Events Committee (CEC) adjudicated.
Time Frame: 6 Months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | SAPIEN THV
Number analyzed (Participants) | 69
percentage of participants | 94.1 [85.1 to 97.8]
Statistical Analysis 1: Comparison: SAPIEN THV; Freedom from Major Adverse Cardiovascular and Cerebrovascular Event (MACCE) at 6 months in the valve implant population; Test type: Superiority or Other; Kaplan-Meier = 0.941, 95% CI 2-sided [0.851 to 0.978], Standard Error of Mean 0.028

3. Secondary Outcome: Functional Improvement
Description: Functional improvement at 6 months as defined by:
  a) Improved valve hemodynamics as demonstrated via Transthoracic Echo: i) Decrease in pulmonary regurgitation to mild or less for regurgitant lesions ii) Decrease in mean pulmonary gradient to less than 30 mmHg for stenotic lesions iii) Improvement in both i) and ii) above for mixed lesions b) Improvement of ≥ 1 NYHA functional class from baseline for patients with NYHA functional class ≥ 2 at baseline c) Freedom from recurrent pulmonary stenosis.
Time Frame: 6 months
Population: Valve implant population. There were 2 screen failure patients and 10 patients where procedure was started but the study valve not implanted, leaving 69 patients in the Valve Implant Population. There were 11 additional patients for which data was not available for analysis, leaving 58 patients in this analysis.
Measure: Number; unit: participants
Arm/Group | SAPIEN THV
Number analyzed (Participants) | 58
participants | 51
Statistical Analysis 1: Comparison: SAPIEN THV; Overall functional improvement at 6 months for patients in the valve implant population with baseline and 6 month data; Test type: Superiority or Other; Percentage = 87.9

ADVERSE EVENTS:
Time Frame: All events.
Description: Site reported.
Arm/Group | SAPIEN THV
Serious Adverse Events (participants affected / at risk) | 38/79
Other Adverse Events (participants affected / at risk) | 47/79
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SAPIEN THV (N=79)
Anemia (Blood and lymphatic system disorders) | 1 (1)
Angina (Cardiac disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 6 (8)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Bleeding Event (Vascular disorders) | 1 (1)
CHF (Cardiac disorders) | 4 (11)
Device migration (Injury, poisoning and procedural complications) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Electrolyte and/or CBC and platelet counts abnormal (Blood and lymphatic system disorders) | 2 (11)
Embolism: air or thrombus (Vascular disorders) | 1 (1)
Endocarditis (Infections and infestations) | 3 (4)
Fever (General disorders) | 4 (4)
Hematoma (Vascular disorders) | 2 (2)
Hemolysis (Blood and lymphatic system disorders) | 1 (1)
Hemorrhage requiring transfusion (Vascular disorders) | 3 (3)
Hemorrhagic event (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Infection (excluding endocarditis) (Infections and infestations) | 7 (12)
Ischemia (Vascular disorders) | 1 (1)
MI (Cardiac disorders) | 1 (1)
Neurological Event (including TIA, stroke and psychomotor deficit) (Nervous system disorders) | 1 (1)
Non-emergent reoperation (Surgical and medical procedures) | 1 (1)
Nonstructural valve dysfunction (Cardiac disorders) | 1 (1)
Pulmonary artery perforation - rupture of RVOT conduit (Injury, poisoning and procedural complications) | 5 (5)
Respiratory complication (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Syncope (Nervous system disorders) | 3 (3)
Thromboembolism (Vascular disorders) | 1 (1)
Valve damage or dysfunction (Cardiac disorders) | 3 (3)
Valve stenosis (Cardiac disorders) | 6 (9)
Other (General disorders) | 13 (37)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SAPIEN THV (N=79)
Anemia (Blood and lymphatic system disorders) | 4 (4)
Angina (Cardiac disorders) | 3 (3)
Arrhythmia (Cardiac disorders) | 8 (10)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Bleeding Event (Vascular disorders) | 9 (10)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Electrolyte and/or CBC and platelet counts abnormal (Blood and lymphatic system disorders) | 5 (5)
Endocarditis (Infections and infestations) | 1 (1)
Fever (General disorders) | 4 (4)
Hematoma (Vascular disorders) | 1 (1)
Hemolysis (Blood and lymphatic system disorders) | 1 (1)
Hemorrhage requiring transfusion (Vascular disorders) | 2 (2)
Hemorrhagic event (Vascular disorders) | 3 (3)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (2)
Infection (excluding endocarditis) (Infections and infestations) | 2 (4)
Neurological Event (including TIA, stroke and psychomotor deficit) (Nervous system disorders) | 1 (1)
Pain at catheterization site (Injury, poisoning and procedural complications) | 2 (2)
Paravalvular leak (Cardiac disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary artery perforation - rupture of RVOT conduit (Injury, poisoning and procedural complications) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory complication (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Syncope (Nervous system disorders) | 3 (4)
Valve damage or dysfunction (Cardiac disorders) | 1 (1)
Valve stenosis (Cardiac disorders) | 1 (1)
Other (General disorders) | 36 (90)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigator will submit to Edwards all manuscripts or presentations authored by investigator and his/her collaborators which result from the Clinical Study at least thirty days prior to submission of the manuscript for publication or presentation.